CLINICAL TRIAL: NCT04477811
Title: Comparative Study Evaluating the Effect of the Administration of Vitamin K1 Versus Vitamin K2 on Vascular Calcification in Dialysis Patients
Brief Title: Comparative Study Evaluating the Effect of Vitamin K1 Versus Vitamin K2 on Vascular Calcification in Dialysis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Farid, clinical professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: vitamin k in dialysis patients
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: End Stage Renal Disease on Dialysis
MeSH Terms: interventions — Vitamin K 1; Vitamin K 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- vitamin k1 (Active Comparator): vitamin k1 will be given 10 mg thrice a week for 3 months
  Interventions: Drug: Vitamin K1
- vitamin k2 (Active Comparator): vitamin k2 (menaquinone) will be given 90 ug per day orally
  Interventions: Drug: Vitamin k2
- placebo (Placebo Comparator): placebo will be given daily per oral for 3 months
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Vitamin K1 — vitamin k1 tablets
  Other Names: Phylloquinone
  Arms: vitamin k1
Drug: Vitamin k2 — vitamin k2 45 ug tablets twice daily
  Other Names: menaquinone
  Arms: vitamin k2
Other: placebo — placebo tablets
  Arms: placebo

SUMMARY:
To evaluate the effect of supplementation of vitamin K2 (menaquinone, MK-7)vs vitamin k1 on circulating levels of calcification regulators and to assess their safety in patients on regular dialysis patients.

DETAILED DESCRIPTION:
Vascular calcification has emerged as an independent risk factor for cardiovascular morbidity and mortality, especially in chronic kidney disease .

It has a predictive value of poor prognoses and clinical outcomes in CKD patients such as overall mortality and even poor arteriovenous graft maturation .

Vitamin K is essential for the activation of matrix Gla protein (MGP), a powerful inhibitor of tissue calcification, functional vitamin K deficiency may contribute to high vascular calcification (VC) burden in haemodialysis patients; this is process in which mineral is pathologically deposited in blood vessels, mainly in large elastic and muscular arteries such as the aorta and the coronary, carotid, and peripheral arteries.

it is Prospective, Randomized,Placebo Controlled Study

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes aged between 18-75 years
2. Patients on HD greater than 3 months at least.
3. Stable clinical condition (no hospitalization in the previous 3 months)

Exclusion Criteria:

1. Hypersensitivity to vitamin k
2. Participant in an another clinical trial within the past 4 weeks.
3. Judged to be unsuitable as a subject by the attending physician.
4. Patients taking warfarin
5. Patients with known intestinal malabsorption
6. Patients with hypercoagulable state

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
change in serum level of Uncarboxylated MGP | change between baseline and after 3 months
  Measuring the change in serum level of Uncarboxylated MGP as a marker for calcification

SECONDARY OUTCOMES:
parathyroid hormone | change between baseline and after 3 months
  measuring change in serum PTH
serum calcium level | change between baseline and after 3 months
  measuring the change in serum calcium level
serum phosphate level | change between baseline and after 3 months
  measuring the change in phosphate level

CONTACTS AND LOCATIONS:
Overall Officials: sarah fahmy, Principal Investigator — Ain Shams University
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palit S, Kendrick J. Vascular calcification in chronic kidney disease: role of disordered mineral metabolism. Curr Pharm Des. 2014;20(37):5829-33. doi: 10.2174/1381612820666140212194926. PMID 24533939
- [Background] McCabe KM, Adams MA, Holden RM. Vitamin K status in chronic kidney disease. Nutrients. 2013 Nov 7;5(11):4390-8. doi: 10.3390/nu5114390. PMID 24212088